CLINICAL TRIAL: NCT02952183
Title: Exploratory Study for Evaluating the Efficacy of Pelvic Autonomic Nerve Monitoring System (PAMS I) in Female Patients With Pelvic Tumors (FUSION Trial V)
Brief Title: Efficacy of Pelvic Autonomic Nerve Monitoring System (PAMS I) in Female Patients With Pelvic Tumors
Acronym: FUSION V
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-2092
Record Dates: First submitted 2016-10-17; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Cervical Cancer; Uterine Cancer; Ovarian Cancer
Keywords: Autonomic nerve monitoring; Nerve-sparing surgery
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PAMS I (Experimental): During operation, autonomic nerve monitoring will be performed by PAMS I which is composed of two urodynamic systems.
  Interventions: Device: PAMS I

INTERVENTIONS:
Device: PAMS I — After general anesthesia, pressure sensor of PAMS I is placed into bladder, vagina and rectum. Then pressure change is monitored during performing pelvic autonomic nerve dissection.
  Both PAMS I and IOM will be used for monitoring.

SUMMARY:
Although nerve-sparing surgery has been introduced for female patients with the pelvic tumors, its success rate depends on operators. To achieve consistency of surgical procedure, It is necessary to adopt pelvic autonomic nerve monitoring technique.

The Aims of this study is

1. Development of pelvic autonomic nerve monitoring system (PAMS I) by using urodynamic system.
2. Evaluation of autonomic nerve sparing by intraoperative monitoring with PAMS I
3. Evaluating the efficacy of PAMS I by intraoperative neurophysiological monitoring (IOM)

DETAILED DESCRIPTION:
After surgery for pelvic tumor, most of patients complain voiding dysfunction, defecation dysfunction and sexual dysfunction which lead to decrease quality of life. Recently, nerve-sparing surgery has been introduced. But it is difficult to establish standard surgical procedure for nerve-sparing. And it is the concern that performing nerve sparing surgery may reduce radicality of surgery which influence prognosis.

Through pelvic autonomic nerve monitoring system (PAMS I), this trial is expected to raise the possibility of nerve-sparing with maintaining radicality of surgery.

Pressure sensor of PAMS I and needle prove of IOM are very thin and these instruments have been used clinically. Taking this into consideration, additional risk by nerve monitoring is considered to be minimal.

ELIGIBILITY:
Inclusion Criteria:

* Female, Age ≥ 18 years
* Patients with pelvic malignant tumor who need surgery.

  * Gynecologic cancer; cervical cancer, uterine cancer, ovarian cancer
  * Colorectal cancer
  * Pelvic sarcoma and metastatic pelvic malignant tumor
* Patients who signed an approved informed consent.

Exclusion Criteria:

* Female, Age < 18 years
* Patients with pelvic malignant tumor, but surgery is not indicated.
* Patients who refused to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Evaluating efficacy of PAMS I by comparison with IOM | Intraoperative
  Comparision pressure change on PAMS I with nerve conduction on IOM
  i) PAMS I (+) & IOM (+): nerve-sparing
  ii) PAMS I (-) & IOM (-): nerve damage
  iii) PAMS I (+) & IOM (-) or PAMS I (-) & IOM (+): intermediate

SECONDARY OUTCOMES:
Evaluation of Quality of life. | Preoperative, 3 months after surgery
  Voiding/Defecation/Sexual function
Time period for recovering normal voiding function | postoperative (up to 6 month)
  Check residual urine. Keep CIC until residual urine < 100cc
Urodynamic test | Preoperative, 3 months after surgery
Anorectal manometry | Preoperative, 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided